CLINICAL TRIAL: NCT04087733
Title: Effectiveness of Liposomial Ozonized-Oil on Ocular Microbial Flora Before Cataract Surgery
Brief Title: Effectiveness of Liposomial Ozonized-Oil for Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Molise (Other)
Collaborators: Azienda Policlinico Umberto I, Roma (Unknown); Università degli Studi del Molise, Clinica Oculistica (Unknown); Clinica Mediterranea, Napoli (Unknown); Ospedale Santa Croce-Carle Cuneo (Other); Centro Medico Oculistico ALSO, Saronno (Unknown); Fondazione G.B. Bietti, IRCCS , Roma (Unknown); Ospedale San Carlo di Nancy, Roma (Unknown); Centro oftalmologico LASERVISTA, Caserta (Unknown); Casa di cura GEPOS, Telese (Unknown); Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other); Ospedale generale regionale F. Miulli, Acquaviva delle Fonti (Unknown); Azienda Ospedaliera Universitaria Mater Domini, Catanzaro (Other); Ospedale Policlinico Casilino, Roma (Unknown); Ospedale G. Panico, Tricase (Unknown); Studio oculistico Laborante (Unknown); Studio oculistico Franchini (Unknown); U.C.O Ospedali Civico di Cristina Benfratelli (Unknown); A.O.U. Città della Salute e della Scienza - Molinette Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0003-08-2018
Record Dates: First submitted 2019-07-18; First posted 2019-09-12 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Ocular Infections
MeSH Terms: conditions — Eye Infections

STUDY DESIGN:
Intervention Model Description: GROUP / TREATED EYE (OZODROP® ): OZODROP® (ozonized oil 0.5% in liposomes) ophthalmic solution, 2 drops 4 times a day. OZODROP® will be instilled in the eye that will have to undergo cataract surgery.
  GROUP / CONTROL EYE: saline solution 2 drops 4 times a day. As a check it will be used the contralateral eye that will not have to undergo cataract surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GROUP / TREATED EYE (Experimental): OZODROP® (ozonized oil 0.5% in liposomes) ophthalmic solution, 2 drops 4 times a day. OZODROP® will be instilled in the eye that will have to undergo cataract surgery.
  Interventions: Drug: OZODROP
- GROUP / CONTROL EYE (No Intervention): Saline solution 2 drops 4 times a day. As a check it will be used the contralateral eye that will not have to undergo cataract surgery.

INTERVENTIONS:
Drug: OZODROP — 3 days before the cataract surgery (T0), two conjunctival swabs will be taken from the patients enrolled in the study, one in the eye to be operated and one in the control eye, who will be kept at a controlled temperature (+ 2 / + 7 ° C) and sent to the laboratory within 24 hours. Than, starting on the day of collection, the patients will instill the OZODROP® eye drops in the eye to be used (2 drops 4 times a day, 1 drop every 4 hours: 9:00 am, 1:00 pm, 5:00 pm: 00, h21: 00), while the contralateral eye will be treated with a saline solution and it will serve as a control. Immediately before the cataract surgery (T3), the patients enrolled in the study will again receive two conjunctival swabs, one in the eye to be operated and one in the control eye. The last OZODROP® instillation will be carried out 10 minutes before the withdrawal. For the microbiological evaluation, the conjunctival swabs taken at T0 and T3 will be sent to the Microbiology laboratory
  Other Names: liposomal ozone-based solution
  Arms: GROUP / TREATED EYE

SUMMARY:
Evaluation of the antimicrobial efficacy of a liposomal ozone-based solution (OZODROP®) , vs placebo in 200 patients undergoing cataract surgery by phacoemulsification .

The clinical trial will last 3 days of treatment per patient. The conjunctival swab will be taken for each of the two eyes (in treatment and control) at T0 (before starting the treatment - 3 days before the cataract surgery) and at T3 (after 3 days of treatment - immediately before the cataract surgery). The last OZODROP instillation will take place 10 minutes before taking the sample.

DETAILED DESCRIPTION:
The aim of the study is to assess the efficacy of a liposomal ozone-based solution (OZODROP®) in the preparation of the patient for cataract surgery, by evaluating the reduction of bacterial colonization of the conjunctiva.

The study will be carried out at 18 surgical centers located throughout the national territory and will be conducted in accordance with the recommendations of Italian ethics committees.

An informed consent will be provided to all study participants. 400 eyes of 200 patients undergoing cataract surgery by phacoemulsification will be included in the study. The clinical sample is divided into two groups, study group which will include treated and (GS) and control group (GC) eyes. The study group will be treated with OZODROP®, an isotonic ophthalmic solution composed of 0.5% ozonized oil in liposomes and hypromellose, while the GC will receive saline solution.

At the time of recruitment, all eyes will undergo a complete examination, as usual, and the patient enrolled in the study will be shown how to proceed.

The study includes 2 times, (T0) and (T3), equal for both groups in the study. 3 days before the cataract surgery (T0), two conjunctival swabs will be taken from the patients enrolled in the study, one in the eye to be operated and one in the control eye, who will be kept at a controlled temperature (+ 2 / + 7 ° C) and sent to the laboratory within 24 hours. Than, starting on the day of collection, the patients will instill the OZODROP® eye drops in the eye to be used (2 drops 4 times a day, 1 drop every 4 hours: 9:00 am, 1:00 pm, 5:00 pm: 00, h21: 00), while the untreated contralateral eye will serve as a control.Immediately before the cataract surgery (T3), the patients enrolled in the study will again receive two conjunctival swabs, one in the eye to be operated and one in the control eye. The last OZODROP® instillation will be carried out 10 minutes before the withdrawal. For the microbiological evaluation, the conjunctival swabs taken at T0 and T3 will be sent to the Microbiology laboratory. The reduction of conjunctival microbial flora, expressed as CFU, will be evaluated.

Through the analysis of the parameters in the study, a significant reduction in the microbial flora of the conjunctiva is expected in patients undergoing treatment with OZODROP®.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years
2. Patients eligible for cataract surgery
3. Willingness to participate in the study following the indications

Exclusion Criteria:

1. Use of topical and / or systemic antibiotics and other topical antiseptics during the study
2. Presence of topical ocular therapies that cannot be suspended for the entire duration of the study
3. Ongoing ocular or systemic inflammatory or infectious processes
4. Hypersensitivity to the constituents of the preparation in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Reduction of conjunctival bacterial load assessed by CFU (Colony Forming Units) using Ozodrop in 200 patients before cataract surgery | 3 days
  Reduction/eradication of conjunctival bacterial load in patients treated with ozodrop for three days before undergoing cataract surgery.
  For the microbiological evaluation, the conjunctival swabs taken at T0 (before starting OZODROP instillation) and T3 (after instilling OZODROP 4 times/day for three days) will be sent to the Microbiology laboratory to be seeded, enriched and then isolated the different species under examination by suitable selective media. The different samples will be analyzed according to the routine methods used in microbiology. The untreated contralateral eye will serve as a control.

CONTACTS AND LOCATIONS:
Overall Officials: Ciro Costagliola, Principal Investigator — University of Molise
Locations (1):
- University of Molise, Campobasso, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Reduction in bacterial load using hypochlorous acid hygiene solution on ocular skin. — https://www.ncbi.nlm.nih.gov/pubmed/28458509
- See also: Human Microbiota and Ophthalmic Disease. — https://www.ncbi.nlm.nih.gov/pubmed/27698616
- See also: Aqueous chlorhexidine (0.1%) is an effective alternative to povidone-iodine for intravitreal injection prophylaxis — https://www.ncbi.nlm.nih.gov/pubmed/26947261
- See also: escrs guidelines — https://www.escrs.org/
- See also: Reduction of anterior chamber contamination rate after cataract surgery by intraoperative surface irrigation with 0.25% povidone-iodine. — http://www.ncbi.nlm.nih.gov/pubmed/20970112
- See also: Sub-Conjunctival Injection of Antibiotics vs. Povidone-Iodine Drop on Bacterial Colonies in Phacoemulsification Cataract Surgery. — http://www.ncbi.nlm.nih.gov/pubmed/25485065
- See also: Study of the Acute Effects of Povidone-Iodine on Conjunctival Bacterial Flora. — http://www.ncbi.nlm.nih.gov/pubmed/26287981
- See also: Evaluation of corneal damage caused by iodine preparations using human corneal epithelial cells. — http://www.ncbi.nlm.nih.gov/pubmed/25230910
- See also: Effect of Povidone Iodine 5% on the Cornea, Vision, and Subjective Comfort. — http://www.ncbi.nlm.nih.gov/pubmed/28609415
- See also: Fourth-generation fluoroquinolones: new topical agents in the war on ocular bacterial infections. — http://www.ncbi.nlm.nih.gov/pubmed/15232471
- See also: Effect of prophylactic antibiotics on antimicrobial resistance of viridans streptococci in the normal flora of cataract surgery patients. — http://www.ncbi.nlm.nih.gov/pubmed/15030817
- See also: Preoperative topical moxifloxacin 0.5% and povidone-iodine 5.0% versus povidone-iodine 5.0% alone to reduce bacterial colonization in the conjunctival sac. — http://www.ncbi.nlm.nih.gov/pubmed/19969216
- See also: Antibacterial activity of ozonized sunflower oil (Oleozon). — http://www.ncbi.nlm.nih.gov/pubmed/11168731
- See also: Ozonated sesame oil enhances cutaneous wound healing in SKH1 mice. — http://www.ncbi.nlm.nih.gov/pubmed/21134039